CLINICAL TRIAL: NCT06032299
Title: Pilot for Dual Implant Versus Single Implant Distal End of Femur (pDISIDE Femur)
Brief Title: Dual Implant Versus Single Implant Distal End of Femur
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brandon James Yuan, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-004415
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Distal Femur Implant Group (Active Comparator): Subjects will receive one of two types of implants for the distal femur fracture. The single implant will be either a plate and screws or a rod. The type of single implant used will be determined by the surgeon based on the characteristics of the fracture.
  Interventions: Procedure: Single Distal Femur Implant
- Dual Distal Femur Implant Group (Experimental): Subjects will receive two implants for fixation of the distal femur fracture. The dual implant will be either 2 plates with screws or a plate with screws and a rod. The type of dual implant used will be determined by the surgeon based on the characteristics of the fracture.
  Interventions: Procedure: Dual Distal Femur Implant

INTERVENTIONS:
Procedure: Single Distal Femur Implant — Single implant constructs will be either a retrograde intramedullary nail with interlocking screws or a single plate and screw construct.
  Arms: Single Distal Femur Implant Group
Procedure: Dual Distal Femur Implant — Dual implant constructs will either be an intramedullary nail with an additional plate and screw construct or dual (two plates in any orientation) plate and screw construct.
  Arms: Dual Distal Femur Implant Group

SUMMARY:
This research study is being conducted to examine the effect of two versus one fixation device for fixation of distal femur fractures.

ELIGIBILITY:
Inclusion Criteria:

* Femur fracture distal to the femoral diaphysis.
* Operative treatment within 72 hours of presenting to the treating hospital.
* Patient was previously ambulatory.
* Fracture amendable to either single or dual implant fixation.
* Informed consent can be obtained from the patient, family member, or power of attorney.

Exclusion Criteria:

* Associated major lower extremity fracture.
* Ongoing infection.
* History of metabolic bone disease (Paget's, etc).
* Pathologic fracture.
* Open fracture.
* Severe cognitive impairment (Six Item Screener with 3 or more errors).
* Stage 5 Parkinson's disease.
* Significant femoral bone loss requiring planned staged bone grafting.
* Vascular injury.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of study-eligible subjects | Baseline
  Total number of subjects to be enrolled in the study

SECONDARY OUTCOMES:
Operative times | Duration of surgery, approximately 2-4 hours
  Total recorded amount of time in minutes to complete the surgery
Blood loss | Duration of surgery, approximately 2-4 hours
  Total amount of surgical blood loss, reported in mL.
Hospitalization days | approximately 2-3 days
  Total number of days a subject requires hospitalization after surgery
Early post-surgical complications | 2 weeks post-surgery
  Number of subjects to experience venous thromboembolism (VTE), cardiopulmonary, and/or infectious complications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Yuan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No